CLINICAL TRIAL: NCT02439008
Title: Early Biomarkers of Tumor Response in High Dose Hypofractionated Radiotherapy Word Package 3 : Immune Response
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient enrollment
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut de Biologie de Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EarlyBio-HypoRT-WP3-1504
Record Dates: First submitted 2015-04-27; First posted 2015-05-08 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Carcinoma, Hepatocellular; Colorectal Neoplasms; Melanoma; Kidney Neoplasms
Keywords: liver metastases of colorectal cancer; metastases of melanoma or renal cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms; Melanoma; Kidney Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood samples collection (Experimental): Nine blood samples will be collected in each patient before, during and after radiotherapy treatment.
  Interventions :
  * Blood samples collection before radiotherapy (T0)
  * Blood samples collection during radiotherapy (T1-T3)
  * Blood samples collection after radiotherapy (T4-T8)
  Interventions: Procedure: Blood samples collection before radiotherapy; Procedure: Blood samples collection during radiotherapy; Procedure: Blood samples collection after radiotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Procedure: Blood samples collection before radiotherapy — Nine blood samples (35 mL each) will be collected in each patient before, during and after radiotherapy treatment.
  Before radiotherapy:
  * Sample T0: after registration, in the days running up to the administration of the first fraction of radiotherapy
Procedure: Blood samples collection during radiotherapy — * Sample T1: within 15 minutes after the administration of the first fraction,
  * Sample T2: within 15 minutes after the administration of the second fraction,
  * Sample T3: within 15 minutes after the administration of the third fraction
Procedure: Blood samples collection after radiotherapy — * Sample T4: one week after the end of the radiotherapy,
  * Samples T5 to T8: respectively 3 months, six months, 9 months and 12 months after the end of the radiotherapy.
Radiation: Radiotherapy

SUMMARY:
This study will follow-up immune cell populations, secreted factors and released nanovesicles in the blood before, during and after high dose radiation therapy which should give new information of the efficacy of the hypofractionated high dose radiation therapy and a rationale for adjuvant immunotherapy.

DETAILED DESCRIPTION:
* Patient information and collection of a signed informed consent form
* Clinical data collection
* Blood samples of 35 mL:

  1. after registration, prior to the first fraction of radiotherapy
  2. within 15 minutes after the administration of the 1st, the 2nd and the 3rd radiotherapy sessions
  3. one week, 3 months, 6 months, 9 months and 12 months after the last radiotherapy session
* Storage of the blood samples at ambient temperature
* Transportation of the samples to the Institute of Biology of Lille (IBL) - CNRS UMR8161 for analysis
* Destruction of the samples at the end of the analysis

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring a hypofractionated irradiation (≥ 3 fractions, dose ≥ 9 Gy per fraction) either for :
* hepatocellular carcinoma or hepatic lesion of metastatic Colorectal Cancer,
* metastasis from melanoma or renal cancer,
* Age ≥ 18 years old,
* Registered with a social security system,
* Signed written informed consent.

Exclusion Criteria:

* Patient treated by chemotherapy, targeted or immunotherapy within 21 days before the first sampling,
* Pregnant or breastfeeding woman,
* Patient under guardianship or tutorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Analyse of immunological parameters, decription of secreted markers and nanovesicles production | from baseline to 1 year follow up
  Description and evolution of cell fraction, quantification of immune cells, verification of the presence and evolution of activation markers and quantification of secreted exosomes ; before, during and after radiotherapy

SECONDARY OUTCOMES:
Cell viability, determined by number of live/dead cells present | from baseline to 1 year follow up
  Cell viability and cell proliferation
Progression-free rate | from baseline to 1 year follow up
  progression-free rate at 12 months
Number of Participants with Adverse Events related to radiotherapy | from baseline to 1 year follow up
  adverse effects (acute toxicity) according to CTCAE-NCI

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mirabel, MD, Study Director — Centre Oscar Lambret; Nadira Delhem, MD, Study Director — Institut de Biologie de Lille
Locations (1):
- Centre Oscar Lambret, Lille, France